CLINICAL TRIAL: NCT06954116
Title: A Prospective, Open-Label, Single-Arm, Exploratory Clinical Study on the Anti-Recurrence Effect of Neoadjuvant Iparomlimab and Tuvonralimab in Resectable Hepatocellular Carcinoma With High Risk of Recurrence After Radical Resection
Brief Title: Iparomlimab and Tuvonralimab as Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma With High Risk of Recurrence
Acronym: CCGLC-017
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ze-yang Ding, MD, Prof., Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202503089
Record Dates: First submitted 2025-04-09; First posted 2025-05-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Resectable Hepatocellular Carcinoma With High Risk of Recurrence
Keywords: Hepatocellular Carcinoma; Neoadjuvant Therapy; Iparomlimab and Tuvonralimab; Immunotherapy; Anti-recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Iparomlimab and Tuvonralimab (Experimental): Patients will receive a single preoperative dose of Iparomlimab and Tuvonralimab (7.5 mg/kg) within one week prior to surgery. Partial hepatectomy will be performed at an appropriate interval following neoadjuvant therapy initiation. From the second week postoperatively, adjuvant therapy with six cycles of Iparomlimab and Tuvonralimab (7.5 mg/kg, Q3W) will be administered.
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706); Procedure: Partial hepatectomy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706) — Neoadjuvant phase: A single cycle of Iparomlimab and Tuvonralimab (7.5 mg/kg) will be administered within 1 week prior to surgery.
  Adjuvant phase: Six cycles of Iparomlimab and Tuvonralimab (7.5 mg/kg, Q3W) will be initiated starting at 2 weeks postoperatively.
Procedure: Partial hepatectomy — Will be performed at an appropriate interval following neoadjuvant therapy initiation.

SUMMARY:
The purpose of this study is to evaluate the impact of iparomlimab and tuvonralimab as preoperative neoadjuvant therapy on recurrence-free survival (RFS), along with its potential improvement in overall survival (OS), in patients with resectable hepatocellular carcinoma (HCC) at high risk of recurrence.

DETAILED DESCRIPTION:
CCGLC-017 is a prospective, open-label, single-arm, exploratory clinical study. This study primarily evaluates the impact of iparomlimab and tuvonralimab (QL1706) as preoperative neoadjuvant therapy on recurrence-free survival (RFS), with exploratory analysis of its potential benefits on overall survival (OS) in patients with resectable hepatocellular carcinoma (HCC) at high risk of recurrence. Enrolled patients will receive a single dose of iparomlimab and tuvonralimab within one week prior to surgery, followed by six cycles of iparomlimab and tuvonralimab therapy postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma is proven on biopsy or confirmed by the presence of radiological hallmarks, according to the American Association for the Study of Liver Diseases or European Association for the Study of the Liver guidelines.
* Aged 18 to 75 years.
* BCLC A/B, or BCLC C without extrahepatic metastasis.
* Suitable for radical surgery after evaluation by the hepatobiliary tumor MDT expert group.
* No distant metastasis confirmed by CT or MRI.
* No prior systemic anti-tumor treatment for hepatocellular carcinoma before the first dose.
* ECOG ≤ 2.
* Child-Pugh ≤ 7.
* Adequate organ and bone marrow function, with laboratory test values meeting the following requirements within 7 days prior to inclusion (no blood components, cell growth factors, albumin, or other intravenous or subcutaneous corrective treatment drugs are allowed within 14 days prior to obtaining laboratory tests):

  1. Complete blood count: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin (HGB) ≥9.0 g/dL.
  2. Liver function: Total Bilirubin (TBIL) ≤2×Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤5×ULN; Serum albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN.

C. Kidney function: Serum Creatinine (Cr) ≤ 1.5×ULN or Clearance of Creatinine (CCr) ≥50mL/min (Cockcroft-Gault formula); Urinalysis shows proteinuria <2+; For subjects with baseline urinalysis showing proteinuria ≥2+, a 24-hour urine collection should be performed and 24-hour urinary protein quantification <1g.

D. Coagulation function: International Normalized Ratio (INR) ≤2.3 or Prothrombin Time (PT) extension ≤6 seconds.

* Meet the criteria for resectable HCC with High Risk of Recurrence:

  1. Multiple (≥2) tumors.
  2. Segmental portal vein invasion (Vp1/Vp2).
  3. CT/MRI imaging: gross classification: type II, III, IV.
* Estimated life expectancy of ≥12 weeks.
* Female subjects of childbearing age or male subjects whose sexual partners are of childbearing age need to take effective contraceptive measures during the entire treatment period and for 6 months after the last medication.
* Signed written informed consent, and able to comply with the visit and related procedures stipulated in the protocol.

Exclusion Criteria:

* Histologically/cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.
* History of hepatic encephalopathy or liver transplantation.
* Clinically symptomatic pleural effusion, ascites, or pericardial effusion requiring drainage. Subjects with only radiologically detected minimal pleural effusion, ascites, or pericardial effusion without symptoms can be enrolled.
* Acute or chronic active hepatitis B or C infection, with hepatitis B virus (HBV) DNA >2000IU/ml or 10^4 copies/ml; hepatitis C virus (HCV) RNA >10^3 copies/ml; co-positive for hepatitis B surface antigen (HbsAg) and anti-HCV antibody. Subjects who meet the above criteria after antiviral treatment with nucleoside analogs can be enrolled.
* History of esophageal or gastric variceal bleeding due to portal hypertension within the past 6 months. Subjects assessed by the investigator to be at high risk of bleeding.
* Any life-threatening bleeding event within the past 3 months, including those requiring blood transfusion, surgery or local treatment, or continuous drug treatment.
* History or current diagnosis of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function, and other lung diseases.
* Active pulmonary tuberculosis, currently receiving anti-tuberculosis treatment, or received anti-tuberculosis treatment within 1 year prior to the first dose.
* Active autoimmune disease requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) is allowed. History of primary immunodeficiency. Patients with only autoantibody positivity need to be confirmed by the investigator whether there is an autoimmune disease.
* History of arterial or venous thromboembolic events within the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other serious thromboembolic events. Exceptions are made for thrombosis formation related to implanted venous infusion ports or catheters, or superficial vein thrombosis that has stabilized after routine anticoagulation treatment. Preventive use of low-dose low molecular weight heparin (such as enoxaparin 40 mg/day) is allowed.
* Continuous use of aspirin (>325 mg/day) or other known platelet function inhibitors such as clopidogrel or ticlopidine for 10 days within 2 weeks prior to the first dose.
* Uncontrolled hypertension, with systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
* Major surgery (craniotomy, thoracotomy, or laparotomy) or unhealed wound, ulcer, or fracture within 4 weeks prior to the first dose. Minor surgical procedures or tissue biopsy within 7 days prior to the first dose, excluding venous puncture for the purpose of intravenous infusion, are excluded.
* Uncontrolled/uncorrectable metabolic disorders or other non-malignant organ diseases or systemic diseases or secondary reactions to cancer, which can lead to higher medical risk and/or uncertainty in survival evaluation, or other conditions judged by the investigator to be unsuitable for enrollment.
* History of gastrointestinal perforation and/or fistula within the previous 6 months, history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | From the date of achieving complete response (CR) after surgery until the date of first documented recurrence or death from any cause, assessed up to 24 months post-surgery.
  The duration will be calculated from the date of achieving complete response (CR) after surgery to the first documented occurrence of intrahepatic or extrahepatic HCC recurrence, or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | from the date of first treatment to the date of death from any cause, assessed up to 5 years
  Overall survival (OS): measured from date of first treatment to the date of death from any cause. Participants alive or lost to follow-up will be censored at the date of their last visit.
Major Pathological Response (MPR) | Intraoperative frozen section assessment and final postoperative pathology (assessed within 4 weeks after surgery).
  Defined as the presence of ≤50% residual viable tumor cells in the resected specimen confirmed by postoperative pathological examination.
Investigator-Assessed Recurrence-Free Survival (RFS) | From treatment initiation until the date of first documented HCC recurrence or death from any cause, whichever occurs first, assessed up to 24 months.
  Defined as the time from treatment initiation to the first documented intrahepatic or extrahepatic HCC recurrence, or death from any cause (whichever occurs first), as determined by the investigator.
Time to Recurrence (TTR) | From treatment initiation until the date of first documented HCC recurrence, assessed up to 24 months.
  Defined as the time from treatment initiation to the first documented intrahepatic or extrahepatic HCC recurrence event.
IRF-Assessed RFS Rate at 12 and 24 Months | At 12 and 24 months post-treatment.
  Defined as the proportion of patients without documented intrahepatic/extrahepatic HCC recurrence or death from any cause at 12 and 24 months post-treatment, assessed by an independent review facility (IRF) using standardized imaging criteria (RECIST 1.1/mRECIST).
Investigator-Assessed RFS Rate at 12 and 24 Months | At 12 and 24 months post-treatment
  Defined as the proportion of patients without documented intrahepatic/extrahepatic HCC recurrence or death from any cause at 12 and 24 months post-treatment, as assessed by the investigator.
OS Rate at 12 and 24 Months | At 12 and 24 months post-treatment initiation.
  Defined as the proportion of patients surviving at 12 and 24 months post-treatment initiation.
Time to Extrahepatic Spread (EHS) or Macrovascular Invasion | From treatment initiation until the date of first documented EHS or macrovascular invasion, assessed up to 24 months.
  Defined as the time from treatment initiation to the first radiologically or histologically confirmed occurrence of either extrahepatic metastasis or macrovascular invasion (portal/hepatic vein involvement).
RFS in PD-L1-High Subgroup or macrovascular invasion (portal/hepatic vein involvement). | From the date of achieving complete response (CR) after surgery until the date of first documented HCC recurrence or death from any cause, whichever comes first, assessed up to 24 months post-surgery.
  Defined as recurrence-free survival in patients with PD-L1-high expression (predefined as combined positive score [CPS] ≥1 by immunohistochemistry) assessed by both investigator and IRF.
Incidence of Adverse Events (AEs) | From the first dose of iparomlimab/tuvonralimab administration until 90 days after the last dose of adjuvant therapy (up to approximately 34 weeks).
  Defined as the proportion of participants experiencing adverse events, graded per Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ze-yang Ding, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China